CLINICAL TRIAL: NCT00644592
Title: LXRA Gene Polymorphisms and Response to Fenofibrate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: supply issues with the formulation of fenofibrate that was used.
Sponsor: University of Florida (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 302-2007
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Results first posted 2012-05-24 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Fenofibrate then Placebo (Active Comparator): 4 weeks of drug at 160 mg orally per day, 4 week washout, then 4 weeks of placebo
  Interventions: Drug: Fenofibrate capsule daily for 4 weeks; Drug: Fenofibrate
- 2 Placebo then Fenofibrate (Active Comparator): 4 weeks of placebo then 4 week washout then 4 weeks of Fenofibrate at 160 mg/day orally.
  Interventions: Drug: Fenofibrate capsule daily for 4 weeks; Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate capsule daily for 4 weeks — Placebo capsule daily for 4 weeks
Drug: Fenofibrate — 160 mg/day orally for 4 weeks

SUMMARY:
This is a research study of how a cholesterol medication known as fenofibrate works differently in people with different genetic backgrounds. "Genetics" refers to certain things that are passed to a person by their parents, such as eye color or hair color. Genetic differences lead to people having different eye and hair color. There are also genetic differences in a protein called liver X receptor-alpha (LXRA), which may be important in predicting the response to fenofibrate.

DETAILED DESCRIPTION:
This is a double blind crossover study of fenofibrate vs. placebo in healthy volunteers. The null hypothesis is that over a four week period, fenofibrate (160mg/day orally) is equivalent to placebo in terms of relative changes in cytokines ENA-78 and MCP-1 over a four week periods, separated by a four week washout. ENA-78 is a marker of inflammation. See http://en.wikipedia.org/wiki/CXCL5 for more details.

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides equal to or above 150mg/dL or Low HDL (below 44 mg/dl for men or below 54 mg/dl for women)
* Must be able to swallow tablets

Exclusion Criteria:

* Known Coronary Heart Disease, symptomatic carotid artery disease, abdominal aortic aneurysm, diabetes, or Framingham risk score above 20%
* Pregnancy, malignancy, liver dysfunction, renal dysfunction, active alcohol abuse, history of unexplained muscle pain
* Current treatment with lipid lowering therapy, estrogens, androgens, progestins, thiazide diuretics, beta-blockers, glucocorticoids (other than inhaled), antihistamines, or chronic anti-inflammatory drugs
* Current treatment with the following the interacting drugs: ursodeoxycholic acid, ursodiol, cholestyramine, red yeast rice, glyburide, glipizide, warfarin, or cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Zineh, PharmD, Principal Investigator — University of Florida College of Pharmacy, Department of Pharmacy Practice, Center for Pharmacogenomics
Locations (1):
- University of Florida College of Pharmacy, Center for Pharmacogenomics, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: UF Clinical Research Center. Started March 2008, completed August 2009.
Pre-assignment Details: Patients were screened for eligibility.
Groups:
- 1-Fenofibrate Then Placebo: 4 weeks of drug at 160 mg orally per day
Period: Overall Study
Arm/Group | 1-Fenofibrate Then Placebo | 2 Placebo Then Fenofibrate
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Fenofibrate Then Placebo | 2 Placebo Then Fenofibrate | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.2 (17.1) | 26.0 (6.6) | 27.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Log(ENA-Period 2 End/ENA Period 1 End)
Description: Log of the ratio of Period end ENA-78 Period 2:Period 1. Once the confidence interval is obtained, we take antilogs to obtain a ratio of effects.
  Natural logs used
Time Frame: week 12 to week 4
Population: Intent was to enroll 30 but drug was withdrawn by provider, with only 11 completing both experimental periods
Measure: Mean (Standard Deviation); unit: Log of Ratio
Arm/Group | 1-Fenofibrate Then Placebo | 2 Placebo Then Fenofibrate
Number analyzed (Participants) | 5 | 6
Log of Ratio | -0.298 (0.31) | 0.178 (0.22)
Statistical Analysis 1: Comparison: 1-Fenofibrate Then Placebo vs 2 Placebo Then Fenofibrate; This is a crossover analysis. To convert to a ratio effect, the mean difference must be divided by two and antilogs take. The outcome represents a relative effect; Test type: Superiority or Other; p = 0.015, t-test, 2 sided; Ratio of mean effects = 1.27, 95% CI 2-sided [1.06 to 1.52], Standard Error of Mean 0.16 — The estimated mean log difference (SE) between the period 2 and period 1 effects and SE was estimated. This estimates twice the effect size[since (B-A)-(A-B)=2B-2A] so the actual estimate was based upon the antilog of half of this difference

ADVERSE EVENTS:
Time Frame: 4 Weeks on Treatment
Groups:
- 1-Fenofibrate: 4 weeks of drug at 160 mg orally per day
- 2 Placebo: 4 weeks of placebo.
Arm/Group | 1-Fenofibrate | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Fenofibrate (N=11) | 2 Placebo (N=11)
Abdominal (Gastrointestinal disorders) | 2 (2) | 0 (0) — Abdominal Complaints
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin rash
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No